CLINICAL TRIAL: NCT06294184
Title: Transcranial Direct Current Stimulation Interventions for Subthreshold Depressive Symptoms in Young Individuals.
Brief Title: TDCS Interventions for Subthreshold Depressive Symptoms in Young Individuals.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Kangguang Lin, Professor, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Guangzhou PH tDCS in SD
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Subthreshold Depression; Young People; Transcranial Direct Current Stimulation
Keywords: Resting-state brain functional network; Social emotion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- lDLPFC tdcs stimulation group (Experimental): The current is 2mA, duration is 1200s, fade in 30s, fade out 30s, anode is on the F3, cathode is on the FP2.
  Interventions: Device: tdcs lDLPFC
- rVLPFC tdcs stimulation group (Experimental): The current is 2mA, duration is 1200s, fade in 30s, fade out 30s, anode is on the F6, cathode is on the FP1.
  Interventions: Device: tdcs rVLPFC
- Sham group (Sham Comparator): The current only persist in the fisrt 30s, duration is 1200s, fade in 30s, fade out 30s, anode is on the F3/F6, cathode is on the FP2/1.
  Interventions: Device: Sham

INTERVENTIONS:
Device: tdcs lDLPFC — The current is 2mA, duration is 1200s, fade in 30s, fade out 30s, anode is on the F3, cathode is on the FP2.
  Arms: lDLPFC tdcs stimulation group
Device: tdcs rVLPFC — The current is 2mA, duration is 1200s, fade in 30s, fade out 30s, anode is on the F6, cathode is on the FP1.
  Arms: rVLPFC tdcs stimulation group
Device: Sham — The current only persist in the fisrt 30s, duration is 1200s, fade in 30s, fade out 30s, anode is on the F3/F6, cathode is on the FP2/1.
  Arms: Sham group

SUMMARY:
The purpose of this study is to assess the mechanisms of the effect of transcranial direct current stimulation (tDCS) in alleviating subthreshold depressive symptoms in young individuals, and individualized outcome prediction is carried out.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all participants providing written informed consent will undergo screening to determine eligibility for study entry. On day 0, participants who meet the eligibility requirements will be randomized in a double-blind manner (participant and investigator) in a 1:1:1 ratio to receive tDCS targeting the left dorsolateral prefrontal cortex (lDLPFC), tDCS targeting the right ventrolateral prefrontal cortex (rVLPFC), or Sham stimulation (10 sessions in 2 weeks). At baseline, after 2 weeks of stimulation, and at follow-up after 1 month and 3 months, participants will be assessed for brain network function, depressive symptoms, emotional status and social interactions.

ELIGIBILITY:
Inclusion Criteria:

* 1) Be between the ages of 12-25;
* 2) is right-handed on the Edinburgh Handedness Inventory;
* 3) 2-4 of the 9 depressive symptoms defined by the American Diagnostic and Statistical Manual of Diseases, Fifth Edition (DSM-5), lasting more than 1 week; or more than 5 depressive symptoms lasting more than 1 week but less than 2 weeks (i.e., not meeting criteria for a major depressive episode) (by DSM-5 Clinical Semi-Definitive Interview (K-SADS-PL) (Gilbody et al., 2017, JAMA);
* 4) Hamilton Depression Scale (HAMD-24) 24 points≥ 8 points, < 24 points;
* 5) Gender is not limited;
* 6) Subjects and their families voluntarily participate and sign the informed consent form.

Exclusion Criteria:

* 1) Individuals with the following diagnoses according to DSM-5: psychiatric disorders due to organic diseases, substance-related and addictive disorders, neurodevelopmental disorders, schizophrenia spectrum and other psychotic disorders, bipolar disorder (assessed by K-SADS-PL);
* 2) Have two or more DSM-V-defined manic symptoms for 4 days but do not meet the criteria for hypomania or meet the DSM-V defined criteria for hypomanic symptoms for only 2-3 days;
* 3) Severe or unstable physical illness;
* 4) have a moderate or higher risk of suicide (as assessed by the Columbia Suicide Severity Scale);
* 5) Received transcranial direct current stimulation in the past three months (continuous intervention time: >2 weeks);
* 6) Contraindications to transcranial direct current stimulation, such as brain implants, personal or family history of epilepsy;
* 7) Magnetic resonance scanning is contraindicated, such as in vivo metal implants.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The effect of tDCS in alleviating subthreshold depressive symptoms | 2 weeks, 1 month and 3 months
  In young individuals with subthreshold depressive symptoms, we used a latent growth model to test whether 10 trials of tDCS for stimulation of lDLPFC or rVLPFC had immediate and sustained (1 & 3 months follow-up) effects on altered depressive symptoms, LPFC-DMN function regulation, positive and negative emotional processing. The latent growth curve model can fit the data well at multiple time points and analyze the correlation of the rate of change of multiple variables. We will measure participants' emotions using the original word score that has been pre-experimentally confirmed, and use the Dynamic Causal Modelling to calculate the resting-state functional regulation of LPFC to DMN (rsFC intensity from LPFC to DMN). We randomized young individuals 1:1:1 to lDLPFC, rVLPFC, and pseudo-stimulation (sham) to test the tDCS effect.

SECONDARY OUTCOMES:
Neuroaffective mechanisms of tDCS in alleviating subthreshold depressive symptoms | 2 weeks, 1 month and 3 months
  We will examine the cross-sectional association between LPFC-DMN functional regulation, positive and negative emotional processing, and depressive symptoms at each time point, and test whether there is a longitudinal association between the immediate and persistent effects of tDCS on the above variables. We will use the cross-lagged structure equation model to test whether the effects of tDCS on LPFC-DMN functional regulation (neural mechanism) and positive and negative emotional processing (affective mechanism) significantly mediate the effect of tDCS on depressive symptoms (outcome variables). We will clarify the temporal sequence of mechanism-outcome effects by testing whether mechanism effects at earlier time points can prospectively predict outcome effects at subsequent time points to infer causal relationships.
To predict the individual effect of tDCS in alleviating subthreshold depressive symptoms | 2 weeks, 1 month and 3 months
  Based on the above analysis results, we will use the Connectome-Based Predictive Model (CPM) method to construct emotional neural data models that predict individual effects. With the advantage of data fitting in machine learning methods, we will screen emotional neurovariables that are significantly related to the level and change of depressive symptoms based on the results of the above mechanism, and build a prediction model around them. We will focus on testing a machine learning model that prospectively predicts the effect of individual interventions: this model will use baseline or earlier time point data to predict the tDCS effect longitudinally at subsequent time points of individual participants. We will also integrate all variables that are cross-sectionally and vertically associated with the level and change of solitary autonomy to build a comprehensive predictive model.

CONTACTS AND LOCATIONS:
Overall Officials: Kangguang Lin, M.D;PH.D, Study Director — The Affiliated Brain Hospital of Guangzhou Medical University; Robin Shao, Ph.D, Principal Investigator — The Affiliated Brain Hospital of Guangzhou Medical University
Locations (1):
- Guangzhou Brain hospital(Guangzhou Huiai Hospital), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No